CLINICAL TRIAL: NCT04150835
Title: Xingnaojing for Mild-to-severe Acute Ischemic Stroke (XMAS-2): A Multicenter, Randomized, Double-blind, Placebo-Controlled Trial
Brief Title: Xingnaojing for Mild-to-severe Acute Ischemic Stroke
Acronym: XMAS-2
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dongzhimen Hospital, Beijing (Other)
Collaborators: Peking University Third Hospital (Other); Beijing Shuyi Hospital (Other); The Airport Hospital of Shunyi District Beijing (Unknown); Cangzhou Hospital of Integrated Traditional Chinese and Western Medicine (Other); The NO.4 People's Hospital of Hengshui (Unknown); The Second Hospital of Hebei Medical University (Other); The Second Affiliated Hospital of Henan University of Traditional Chinese Medicine (Other); The Affiliated Hospital of Shaanxi University of Chinese Medicine (Unknown); Tianshui Hospital of Traditional Chinese Medicine (Unknown); The Affiliated Hospital of Changzhi Academy of TCM (Unknown); Zibo Hospital of Traditional Chinese Medicine (Other); Yantai Yuhuangding Hospital (Other); Shandong University of Traditional Chinese Medicine (Other); Zhejiang Provincial Hospital of TCM (Other); Zhejiang Provincial Tongde Hospital (Other); Second Affiliated Hospital of Wenzhou Medical University (Other); People's Hospital of Quzhou (Other); Longhua Hospital (Other); The First Affiliated Hospital of Anhui University of Traditional Chinese Medicine (Other); Taizhou Hospital of Traditional Chinese Medicine (Other Government); The First Affiliated Hospital of Guizhou University of TCM (Unknown); Guangzhou Hospital of Traditional Chinese Medicine (Unknown); The First Affiliated Hospital of Guangxi University of Chinese Medicine (Unknown); Liling Hospital of Traditional Chinese Medicine (Unknown); Hunan Academy of Traditional Chinese Medicine Affiliated Hospital (Unknown); Hubei Hospital of Traditional Chinese Medicine (Other); The First Hospital of Jilin University (Other); Anshan Central Hospital (Other); Affiliated Hospital of Liaoning University of Traditional Chinese Medicine (Other); The First Hospital of Qiqihar City (Unknown); Haikou People's Hospital (Other); The Second People's Hospital of Anhui Province (Other); The Third Affiliated Hospital of Shenzhen University (Unknown); The Third People's Hospital of Hubei Province (Other); The First Affiliated Hospital of Henan University of Traditional Chinese Medicine (Other); The Third Hospital of Xi'an City (Unknown)
Responsible Party: Principal Investigator, Ying Gao, President of the Institute for Encephalopathy, Beijing University of Chinese Medicine, Dongzhimen Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018YFC1705001
Record Dates: First submitted 2019-11-01; First posted 2019-11-05 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Acute Ischemic Stroke; Stroke, Acute; Stroke, Ischemic
Keywords: Acute ischemic stroke; Xingnaojing injection; Traditional Chinese Medicine; Double-Blind; Randomized Controlled Trial
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — xingnaojing; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Xingnaojing (Experimental): Subjects will receive intravenously administered Xingnaojing injection, combined with guidelines-based standard care.
  Interventions: Drug: Xingnaojing injection; Other: Standard care
- Placebo (Placebo Comparator): Subjects will receive intravenously administered Xingnaojing placebo, combined with guidelines-based standard care.
  Interventions: Drug: Xingnaojing placebo injection; Other: Standard care

INTERVENTIONS:
Drug: Xingnaojing injection — Xingnaojing injection (20 ml)+0.9% diluted sodium chloride injection 250ml, IV (in the vein), every 12 hours for 10 days.
  Arms: Xingnaojing
Drug: Xingnaojing placebo injection — Xingnaojing placebo injection (20 ml)+0.9% diluted sodium chloride injection 250ml, IV (in the vein), every 12 hours for 10 days.
  Arms: Placebo
Other: Standard care — Guidelines-based standard care for acute ischemic stroke.

SUMMARY:
The main purpose of this trial is to determine whether Xingnaojing, intravenously administered within 24 hours of symptom onset, improves the daily living ability of acute ischemic stroke at 90 days.

DETAILED DESCRIPTION:
The XMAS-2 study is a multicenter, randomized, double-blind, placebo-controlled clinical trial. The primary hypothesis of this trial is that Xingnaojing will improve the daily living ability of acute ischemic stroke at 90 days. Xingnaojing will be compared to placebo, combined with guidelines-based standard care in patients with acute ischemic stroke within 24 hours of symptom onset. All participants will have a National Institutes of Health Stroke Scale(NIHSS)entry score of 4-25. Participants who have planned or already received the intravenous thrombolysis or endovascular treatment will be excluded. The primary outcome will be determined at 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Acute ischemic stroke；
* Symptom onset within 24 hours；
* Age ≥ 18 and ≤ 80 years；
* NIHSS score ≥ 4 and ≤ 25；
* Patient or legally authorized representative has signed informed consent.

Exclusion Criteria:

* Planned or already receiving intravenous thrombolysis or endovascular treatment;
* Suspected secondary stroke caused by tumor, brain trauma, or hematological diseases;
* Already dependent in activities of daily living before the present acute stroke (defined as modified Rankin Scale score ≥ 2) ;
* Other conditions that cause cardiogenic embolism (e.g., atrial fibrillation, rheumatic heart disease, valvular heart disease);
* Other conditions that lead to motor dysfunction (e.g., severe osteoarthrosis, rheumatoid arthritis);
* Significant renal or hepatic insufficiency (defined as a serum creatinine concentration, alanine aminotransferase (ALT), or aspartate aminotransferase (AST) value that is twice the upper limit of normal);
* Life expectancy of 3 months or less due to other life-threatening illness (e.g.,advanced cancer)
* Other conditions that render outcomes or follow-up unlikely to be assessed;
* Known to be pregnant or breastfeeding;
* Currently receiving an investigational drug;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2020-03-19 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients independent. | 90 days
  Proportion of patients independent is defined as Modified Rankin Scale score of 0, 1, or 2.The Modified Rankin Scale Score ranges from 0 (best score) to 6 (worst score).

SECONDARY OUTCOMES:
Early neurological deterioration. | Baseline and 3 days
  The early neurologic deterioration is defined as an increase of 1 points or more in the National Institute of Health Stroke Scale (NIHSS) score between baseline and 3 days. The NIHSS score ranges from 0 (best score) to 42 (worst score).
Neurological impairment evaluated by National Institute of Health Stroke Scale (NIHSS). | Baseline and 10 days
  Comparison of the change in the NIHSS scores from baseline to 10 days in the two groups.The NIHSS score ranges from 0 (best score) to 42 (worst score).
Patient reported outcome | 10 days
  Patient reported outcome (PRO) scale of stroke at 10 days.The PRO score ranges from 36(best score) to 180 (worst score).
State of consciousness | 48 hours and 7 days
  The state of consciousness evaluated by Glasgow Coma Scale at 7 days. The Glasgow score ranges from 3(worst score) to 15 (best score).
Activities of daily living | 30 days and 90 days
  Activities of daily living will be measured by Barthel Index score at 30 days and 90 days.The Barthel Index score ranges from 0 (worst score) to 100 (best score).
The proportion of patients independent at 30 days. | 30 days
  The proportion of patients independent will be evaluated by mRS at 30 days.The mRS score ranges from 0 (best score) to 6 (worst score).
The recurrence rate of cerebrovascular events | Within 90 days
  The recurrence rate of cerebrovascular events within 90 days.
Stroke related deaths and deaths from any cause | Within 10 days and 90 days
  Stroke related deaths and deaths from any cause within 10 days and 90 days after symptom onset.
Safety end points | 10 days
  Number of patients with any adverse events, results of electrocardiography, vital signs and laboratory tests (complete blood count, chemistry and urinalysis).

CONTACTS AND LOCATIONS:
Overall Officials: Ying Gao, MD, Principal Investigator — Dongzhimen Hospital
Locations (1):
- Dongzhimen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided